CLINICAL TRIAL: NCT07171268
Title: A Randomized Controlled Trial of Yoga Asana Chandra Harmoni on Psychological Well-being and Learning Readiness Among Medical Students
Brief Title: Yoga Asana Chandra Harmoni on Psychological Well-being and Learning Readiness Among Medical Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Made Satya Nugraha Gautama, Principal Investigator, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 025UN481604
Record Dates: First submitted 2025-09-04; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Yoga; Yoga Exercises; Well Being; Self Efficacy; Medical Student; Health and Wellness

STUDY DESIGN:
Intervention Model Description: The Yoga Asana Chandra Harmoni intervention is a structured yoga program based on a specific sequence of asanas, pranayama (breathing exercises), and meditation techniques. The core asana sequence includes both static and dynamic movements designed to promote physical flexibility, strength, and balance. Pranayama techniques focus on regulating the breath to calm the nervous system and reduce stress. Meditation practices aim to cultivate mindfulness and improve emotional regulation. The intervention will be delivered in two phases: an initial face-to-face instruction session, followed by independent practice supported by a video and WhatsApp support. Participants in the intervention group will also be prescribed with online audio guided practices 5 times/week for 20-30 minutes. The audio practice will include breathing exercises (weeks 1-2) and body scans (weeks 3-4).
Who Masked: Outcomes Assessor
Masking Description: To minimize bias, this study will implement masking procedures. Specifically, investigators involved in direct participant interaction will not be masked because of the nature of intervention (yoga classes require a known instructor), The outcome assessors responsible for administering and scoring the questionnaires (DASS-21, PSQI, SDLR, and Self-Efficacy) will be masked to the participant's group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants randomized to the control group will continue with their usual daily activities and academic routines. They will not receive the Yoga Asana Chandra Harmoni intervention during the study period.
  Interventions: Behavioral: Yoga Asana Chandra Harmoni
- Wait-List Control Group (No Intervention): Participants randomized to the wait-list control group will continue with their usual daily activities and academic routines. They will not receive the Yoga Asana Chandra Harmoni intervention during the study period.

INTERVENTIONS:
Behavioral: Yoga Asana Chandra Harmoni — Description: Participants randomized to the intervention group will receive the Yoga Asana Chandra Harmoni program. This program is designed to improve psychological well-being, sleep quality, and self-directed learning readiness.
  Components:
  Initial Face-to-Face Session: Participants will attend one in-person session led by a qualified yoga instructor. This session will introduce the principles of Yoga Asana Chandra Harmoni and provide instruction on the core asana sequence, breathing techniques (pranayama), and meditation.
  Weekly Yoga Sessions: Participants will engage in three 45-minute yoga sessions per week for four weeks, practicing the Yoga Asana Chandra Harmoni sequence.
  Video Support: Participants will be provided with a video demonstrating the Yoga Asana Chandra Harmoni sequence to support their home practice. The video will be shared individually via Whatsapp.
  Home Practice: Participants are expected to practice the Yoga Asana Chandra Harmoni sequence independently at home,
  Arms: Control Group

SUMMARY:
The goal of this trial is to learn if the Yoga Asana Chandra Harmoni intervention can improve psychological well-being and learning readiness in medical students. The main questions it aims to answer are:

Does Yoga Asana Chandra Harmoni improve psychological well-being (specifically, reduce stress, anxiety, and depression) in medical students? Does Yoga Asana Chandra Harmoni enhance self-directed learning readiness in medical students? Researchers will compare a group receiving the Yoga Asana Chandra Harmoni intervention to a control group to see if the intervention leads to significant improvements in psychological well-being and self-directed learning readiness.

Participants will:

Complete baseline questionnaires assessing psychological well-being, sleep quality, self-directed learning readiness, and self-efficacy.

Participate in 3 weekly Yoga Asana Chandra Harmoni sessions for 4 weeks (intervention group).

Continue with their usual activities (control group). Complete follow-up questionnaires at post-test (end of week 4) and at a 2-week follow-up to assess changes in the outcome measures.

Engage in additional online audio guided practices 5 times/week for 20-30 minutes, including breathing exercises (weeks 1-2) and body scans (weeks 3-4) (intervention group).

DETAILED DESCRIPTION:
Background & Rationale

Medical students face significant academic pressures, leading to elevated levels of stress, anxiety, and depression. These psychological challenges can negatively impact their academic performance, sleep quality, and overall well-being. Furthermore, the demands of medical education necessitate effective self-directed learning skills. Yoga interventions have demonstrated potential for improving mental health and cognitive function in various populations. This study aims to rigorously evaluate the effectiveness of a specific yoga intervention, Yoga Asana Chandra Harmoni, in addressing these challenges within a medical student population.

Intervention Details:

The Yoga Asana Chandra Harmoni intervention is a structured yoga program based on a specific sequence of asanas, pranayama (breathing exercises), and meditation techniques. The core asana sequence includes both static and dynamic movements designed to promote physical flexibility, strength, and balance. Pranayama techniques focus on regulating the breath to calm the nervous system and reduce stress. Meditation practices aim to cultivate mindfulness and improve emotional regulation. The intervention will be delivered in two phases: an initial face-to-face instruction session, followed by independent practice supported by a video and WhatsApp support. Participants in the intervention group will also be prescribed with online audio guided practices 5 times/week for 20-30 minutes. The audio practice will include breathing exercises (weeks 1-2) and body scans (weeks 3-4).

Study Design and Procedures:

This study will utilize a randomized controlled trial (RCT) design. Eligible participants will be randomly assigned to either the Yoga Asana Chandra Harmoni intervention group or a control group receiving no intervention. Randomization will be performed using computer-generated random numbers. To ensure minimal contamination, participants will be encouraged not to discuss the intervention with those in the control group.

Adherence to the intervention will be monitored through self-reported practice logs. Participants will be asked to record the frequency and duration of their yoga practice. In the event of significant non-adherence, strategies will be employed to encourage participation, such as reminder messages.

ELIGIBILITY:
Inclusion Criteria:

* 3rd-year medical student
* Willing to attend yoga sessions and practice at home.
* Willing to provide consent and complete assessments.

Exclusion Criteria:

* Regular yoga practice (≥ 6 months).
* Physical contraindications to yoga.
* Active treatment for severe mental health disorder.
* Concurrent participation in another intervention study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Psychological well-being (measured by the Depression Anxiety Stress Scales - DASS-21) | Baseline (Prior to the intervention); Post-test (Immediately following the 4-week intervention period); Follow-up (Two weeks after the post-test assessment).
  The DASS-21 is a self-report instrument that assesses the severity of symptoms of depression, anxiety, and stress experienced by individuals.

SECONDARY OUTCOMES:
Sleep Quality (Measured by the Pittsburgh Sleep Quality Index - PSQI) | Baseline (Prior to the intervention); Post-test (Immediately following the 4-week intervention period); Follow-up (Two weeks after the post-test assessment).
  The PSQI is a self-report questionnaire designed to assess sleep quality and disturbances over a 1-month time interval.
SDLR (measured by the Indonesian version of the Self-Directed Learning Readiness Scale - SDLR) | Baseline (Prior to the intervention); Post-test (Immediately following the 4-week intervention period); Follow-up (Two weeks after the post-test assessment).
  SDLR scale measures an individual's preparedness to engage in self-directed learning activities.
Self-Efficacy (Measured by the Indonesian version of the Student Self-Efficacy Scale) | Baseline (Prior to the intervention); Post-test (Immediately following the 4-week intervention period); Follow-up (Two weeks after the post-test assessment).
  Self-Efficacy scale measures students' belief in their ability to succeed in specific situations or accomplish a task

CONTACTS AND LOCATIONS:
Overall Officials: Made Kurnia Widiastuti Giri, Dr., Principal Investigator — Universitas Pendidikan Ganesha
Locations (1):
- Universitas Pendidikan Ganesha, Singaraja, Bali, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maity S, Abbaspour R, Bandelow S, Pahwa S, Alahdadi T, Shah S, Chhetri P, Jha AK, Nauhria S, Nath R, Nayak N, Nauhria S. The psychosomatic impact of Yoga in medical education: a systematic review and meta-analysis. Med Educ Online. 2024 Dec 31;29(1):2364486. doi: 10.1080/10872981.2024.2364486. Epub 2024 Jun 11. PMID 38861675